CLINICAL TRIAL: NCT07135960
Title: Breast Cancer BRAs Study (Breast Cancer Biomechanics of Radiotherapy And Surgery): The Effects of Breast Surgery and Radiotherapy on the Breast Biomechanics and Breast Support Requirements of Women Treated for Breast Cancer.
Brief Title: Breast Cancer BRAs Study (Breast Cancer Biomechanics of Radiotherapy And Surgery)
Status: Recruiting | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: University of Portsmouth (Other)
Responsible Party: Sponsor
Other Study IDs: PHU/2024/32
Record Dates: First submitted 2025-05-27; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants with relevant condition
- Women aged 18 or treated with surgery +/- radiotherapy for breast cancer that affects one of their b

SUMMARY:
This study, delivered by Portsmouth Hospitals University NHS Trust in conjunction with the Research Group in Breast Health at the University of Portsmouth [1], aims to assess whether it is possible to test breast biomechanics in women who have had surgery with or without radiotherapy for the treatment of breast cancer.

DETAILED DESCRIPTION:
Breast cancer is an increasingly common condition, affecting >56,000 women a year in the UK. Surgery and radiotherapy are commonly used to treat breast cancer. Both these treatments can affect the structure and movement of the breast tissue, which is collectively called breast biomechanics. Breast biomechanics has been studied in healthy women and in female athletes, and across the menstrual cycle, menopause and pregnancy. Investigators know from this research that breast biomechanics can affect the type of bra support women need, which when optimised can improve comfort and quality of life as well as reduce the potential for tissue damage. However, breast biomechanics and associated breast garment support requirements (bra support) have not yet been significantly investigated in women undergoing breast cancer treatment.

Patients who would be eligible to participate in this study include women aged 18 or treated with surgery +/- radiotherapy for breast cancer that affects one of their breasts. Patients will be recruited from the Breast Unit at Queen Alexandra Hospital, Cosham. Participation in this study will involve attending the biomechanics testing laboratory at UoP after their surgery and/or after radiotherapy, and optionally before surgery too. 3D scans and sensors will be used to assess the structure and movement of the breast. Participants will be asked their views on the testing methods, as well as their bra requirements and exercise habits before and after breast cancer treatment. The information generated from this study could be used in the future to help design better bras for women treated for breast cancer. It could also help women make decisions about treatment based on evidence about how the breast is likely to move differently afterwards and improve satisfaction with treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or above
* Early or locally advanced breast cancer classified as B5a or B5b (radical treatment intent)
* Unilateral breast cancer (contralateral breast used as control)
* Receiving or has received breast cancer surgery
* +/- Adjuvant radiotherapy
* Able to travel to the University of Portsmouth Breast biomechanics laboratory
* Participant has capacity to consent.

Exclusion Criteria:

* Metastatic breast cancer diagnosis
* < 2 weeks post-operative
* < 4 weeks post-radiotherapy
* Active post-operative breast infection
* Requirement of ongoing breast dressings
* Previous breast surgery to contralateral breast
* Bilateral breast cancer
* Epilepsy (due to strobe on 3D scanner)
* Pregnancy or <6 weeks post-partum
* Breastfeeding
* Rockwood Frailty score >5 (or those unable to ambulate un-aided)
* Requiring interpreter.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants biological born female
Study Population: Female patients, aged >18, who have a diagnosis of early breast cancer, and are offered breast surgery +/- adjuvant radiotherapy as part of their breast cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
To determine the feasibility of recruitment to a breast biomechanics study in women treated for early breast cancer with surgery +/- adjuvant radiotherapy. | From enrollment to the end of study [through study completion, an average of 1 year]
  To identify:
  Number of patients eligible. Number of patients approached. Number of patients who give informed consent. Number of patients who withdraw after consent before participation. Number of patients who withdraw during follow-up. Number of patients lost to follow-up. Completeness of data per participant. Barriers to participation

SECONDARY OUTCOMES:
To determine if it is possible to obtain breast biomechanics data in women treated for early breast cancer with surgery +/- adjuvant radiotherapy. | From enrollment to the end of study [through study completion, an average of 1 year]
  To collect quantitative data on breast biomechanics.
  To assess:
  Sensitivity of data collection methods to detect differences in breast biomechanics pre-operatively to post-operatively and/or between left breast and right breast.

CONTACTS AND LOCATIONS:
Overall Officials: Edward St John, Principal Investigator — Portsmouth Hospitals University NHS Trust
Locations (1):
- Queen Alexandra Hospital, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No